CLINICAL TRIAL: NCT04300114
Title: A Phase III, Randomised, Double Blind, Placebo Controlled, Multicentre Study of Maintenance Fluzoparib Monotherapy in Patients With gBRCA/PALB2 Mutated Metastatic Pancreatic Cancer Whose Disease Has Not Progressed on First Line Platinum Based Chemotherapy
Brief Title: A Study of Maintenance Treatment With Fluzoparib in gBRCA/PALB2 Mutated Pancreatic Cancer Whose Disease Has Not Progressed on First Line Platinum-Based Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR3162-III-304
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance Fluzoparib monotherapy (Experimental)
  Interventions: Drug: Fluzoparib
- Maintenance placebo monotherapy (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib capsules po. 150 mg twice daily
  Other Names: SHR3162
  Arms: Maintenance Fluzoparib monotherapy
Drug: Placebo — Placebo capsules po. twice daily
  Arms: Maintenance placebo monotherapy

SUMMARY:
The study is being conducted to evaluate the tolerability, safety and efficacy of maintenance Fluzoparib monotherapy in patients with gBRCA/PALB2 mutated metastatic pancreatic cancer whose disease has not progressed on first line platinum based chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Expected survival ≥ 3 months.
* Histologically or cytologically confirmed metastatic pancreas adenocarcinoma.
* Patients who have received a minimum of 16 weeks of continuous platinum treatment for metastatic disease and have no evidence of progression based on investigator's opinion.
* Patients with measurable disease and/or non-measurable or no evidence of disease assessed at baseline by CT or MRI.
* Documented mutation in germline BRCA1/2 or PALB2 that is predicted to be deleterious or suspected deleterious.
* Adequate organ performance based on laboratory blood tests.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Major Exclusion Criteria:

* Previous treatment with a poly ADP-ribose polymerase (PARP) inhibitor.
* Patients who have had radiotherapy within 2 weeks or participated in another clinical trial with any investigational agents within 2 weeks prior to study screening.
* Previous treatment using CYP3A4 inducers within 3 weeks or inhibitors within 2 weeks.
* Significant cardiovascular disease such as New York Heart Associate Class III/IV, cardiac failure, myocardial infarction, unstable arrhythmia, or evidence of ischemia on ECG within 6 months prior to enrolment.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia.
* Known active hepatitis B or C infection.
* History of immunodeficiency (including HIV infection) or organ transplantation.
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
PFS by Blinded Independent Central Review (BICR) Using RECIST v1.1 | up to 3 years
  Progression-Free-Survival

SECONDARY OUTCOMES:
ORR by BICR Using RECIST v1.1 | up to 3 years
  Objective Response Rate
DCR by BICR Using RECIST v1.1 | up to 3 years
  Disease Control Rate
DoR by BICR Using RECIST v1.1 | up to 3 years
  Duration of Response
PFS by Investigators Using RECIST v1.1 | up to 3 years
  Progression-Free-Survival
ORR by Investigators Using RECIST v1.1 | up to 3 years
  Objective Response Rate
DCR by Investigators Using RECIST v1.1 | up to 3 years
  Disease Control Rate
DoR by Investigators Using RECIST v1.1 | up to 3 years
  Duration of Response
OS | up to 3 years
  Overall-Survival
Number of participants with treatment-emergent adverse events | From the first drug administration to within 30 days for the last drug dose
  The number and proportion of subjects experiencing treatment-emergent adverse events (TEAE)

CONTACTS AND LOCATIONS:
Overall Officials: Yupei Zhao, Ph.D, Principal Investigator — Peking Union Medical College Hospital
Locations (23):
- China (23):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The 3rd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shandong Cancer Hospital and Institute, Jinan, Shandon
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affilited to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital Institute, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang